CLINICAL TRIAL: NCT04932226
Title: Peripheral Oxygen Saturations Among Healthy Young Adults Wearing Face Masks Whilst Exercising
Brief Title: Face Masks and Oxygen Levels - What Happens During Exercise? (Masks in Exercise - a RandomIsed Trial)
Acronym: MERIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Nottingham (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PHC_facemasks&exercise1
Record Dates: First submitted 2021-06-17; First posted 2021-06-21 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2021-06

CONDITIONS: Impact of Masks on Oxygen Levels

STUDY DESIGN:
Intervention Model Description: Each participant is own control. Each participant will undergo all four interventions in random order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Other): Each participant is his/her own control. Each will have all four interventions in random order.
  Interventions: Device: cloth mask; Device: surgical mask; Device: FFP2 respirator

INTERVENTIONS:
Device: cloth mask — Buff bandana double layer worn over nose and mouth
Device: surgical mask — standard surgical mask
Device: FFP2 respirator — filtering facepiece 2 respirator

SUMMARY:
The investigators aim to determine the effect of three different types of face mask compared to no face mask on the oxygen saturations, heart rate and symptoms of healthy young adults during 15 minutes of moderate to high intensity exercise. The three face masks will be a cloth mask, a surgical mask and a FFR.

DETAILED DESCRIPTION:
The investigators will conduct a crossover study comparing three different types of face mask (cloth, surgical or filtering facepiece respirator - FFR) versus no face mask to determine the effect on oxygen saturations, heart rate and symptoms of healthy young adults during 15 minutes of moderate to high intensity exercise. The investigators will promote the study through sports societies at three leading United Kingdom (UK) universities, namely the University of Oxford, University of Nottingham and King's College London. The investigators will also advertise the study on social media.

Interested individuals will be encouraged to visit the study website or read the patient information sheets available to share via email. Volunteer participants will be asked to read the eligibility criteria, patient information sheet and recruitment information before applying to take part. Those who wish to participate will be asked to complete an online form, including their first name, date of birth, address, email address, demographics, details of their regular exercise and details of any past medical history or medication.

Those wishing to discuss the study will have the opportunity to request a phone call from a member of the study team before agreeing to take part.

Submitted applications will be screened by the study team for eligibility. Those who are deemed not to be eligible will be contacted, explaining the reason. Selected participants will be informed and contacted to arrange a date for the study session. This will be conducted at their local university sports centre or a local park. The number of participants attending a single study session will be in compliance with any UK government restrictions relating to COVID-19 in place at that time.

On the day of the study, participants will meet a member of the study team, who will ask them to complete an online consent form.

Participants will then be asked to complete an exercise study session. The type of exercise will be either:

* Running
* Cycling
* Rowing on a fixed machine

Participants will be asked to complete four x 15 minute pieces of exercise within this single session. The aim will be to exercise at moderate to high intensity with the goal of covering the same distance each time. Between 15 minutes of exercise, participants will be asked to take a 5 minute rest break. For each 15 minute session, participants will wear one of the following:

* a cloth mask
* a surgical mask
* a FFR
* no mask

The order in which participants wear the face masks will be determined by a random sequence generator(https://www.phc.ox.ac.uk/research/technology-outputs/sortition-clinical-trial-randomisation-software). The masks will be provided by the researcher at the time.

Participants will wear no mask during each rest period. Prior to starting, participants will have their resting heart rate and oxygen levels recorded. Halfway through each exercise period, immediately on completing the exercise and at 1 minute following completion of the exercise, participants will have their heart rate, oxygen levels and distance travelled recorded by a member of the study team.

Upon completion of the exercise session, participants will be asked to complete an online survey via a secure portal, hosted by the University of Oxford. They will be asked to complete questions regarding the type of exercise they did, oxygen levels and heart rate at each time point, distance travelled and average speed, and questions regarding the ease of exercise and comfort of wearing each masks, as well as any additional symptoms they might have experienced during the exercise session as a result of wearing the mask.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 - 35 years old.
* Exercise at least three times a week on a regular basis.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Known to have a significant acute or longstanding medical illness that limits their exercise capacity.
* Develop symptoms of anosmia, cough or fever between agreeing to participate and completing the exercise, suggesting they may have developed COVID-19.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-06-19 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | Immediately after exercise
  Oxygen saturation using pulse oximeter

SECONDARY OUTCOMES:
heart rate | immediately after exercise
  Heart rate
distance traveled | immediately after exercise
  distance traveled as a % of distance traveled when unmasked
comfort | immediately after exercise
  symptom survey of mask comfort and any adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- Trisha Greenhalgh, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Will be placed on a website
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months
Access Criteria: Contact lead author

REFERENCES:
- [Derived] Jones N, Oke J, Marsh S, Nikbin K, Bowley J, Dijkstra HP, Hobbs FR, Greenhalgh T. Face masks while exercising trial (MERIT): a cross-over randomised controlled study. BMJ Open. 2023 Jan 5;13(1):e063014. doi: 10.1136/bmjopen-2022-063014. PMID 36604128